CLINICAL TRIAL: NCT00216502
Title: Long Term Treatment With Galantamine In Dementia
Brief Title: A Study of the Safety and Effectiveness of Galantamine in Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag S.p.A. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004996
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Alzheimer Disease; Dementia; Mental Disorders; Brain Diseases
Keywords: Alzheimer's disease; Dementia; galantamine; placebo; Caregiver; Brain disease; Memory loss
MeSH Terms: conditions — Alzheimer Disease; Dementia; Mental Disorders; Brain Diseases; Memory Disorders | interventions — Galantamine

INTERVENTIONS:
Drug: galantamine hydrobromide

SUMMARY:
The purpose of this study is to evaluate the long-term efficacy and safety of galantamine in patients with Alzheimer's disease.

DETAILED DESCRIPTION:
Dementia is a chronic, progressive brain disease that may involve a number of symptoms, including memory loss and changes in personality, behavior, judgment, attention span, language and thought. The most common type of dementia is Alzheimer's disease. Over time, patients with Alzheimer's disease may lose ability to perform daily tasks related to personal care (for example bathing, dressing, eating) and may be unable to handle money or travel to familiar places. Previous short-term studies have shown galantamine to be safe and effective in treating patients with Alzheimer's disease, however the long-term safety and effectiveness of galantamine have not been examined. This multicenter, randomized study will assess whether long-term treatment with galantamine will delay the onset of symptoms associated with Alzheimer's disease and examine the safety and effectiveness of long-term treatment with galantamine. Patients will receive 12 months of open-label treatment with galantamine, followed by 24 months of double-blind treatment with galantamine or placebo. Safety evaluations (incidence of adverse events, physical examinations, 12 lead ECGs, vital signs, laboratory tests) will be performed throughout the study. Effectiveness will be determined using standard tests and rating scales to assess mental status, functioning, thinking, behavior, judgment and language (Mini Mental Status Exam [MMSE], Alzheimer's Disease Assessment Scale [ADAS-cog]; Disability Assessment for Dementia [DAD], and Clinician's Interview Based Impression of Changes plus Family Input [CIBIC-plus]). After the first 4 weeks, assessments will be performed every 3 months during the open-label phase (first 12 months) and then every 6 months during the double-blind phase (13-36 months). Patients whose symptoms worsen as defined by an increase of > or = to 4 points in their ADAS-cog score from the start of the double-blind phase will be withdrawn from the study. The study hypothesis is that long-term treatment with galantamine will be effective in delaying the cognitive deterioration in patients with Alzheimer's disease and that galantamine is well-tolerated with long term treatment. Galantamine 4 milligrams twice daily by mouth for 4 weeks, then 8 milligrams twice daily for 48 weeks. Thereafter, galantamine will be given as 8 milligrams twice daily for an additional 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer's disease according to accepted medical standards
* Patients with mild to moderate impairment of thinking, reasoning, and judgment as defined by a score from 11-24 on the Mini Mental Status Exam (MMSE, a standard assessment tool for Alzheimer's disease) Female patients must be post-menopausal
* Patients and their caregivers must have signed informed consent forms Exclusion Criteria:
* Patients with a diagnosis of Parkinson's Disease, Pick's Disease, Huntington's Chorea, Creutzfeld-Jacob disease, Down's syndrome, brain cancer, mental retardation, epilepsy, psychiatric disease, liver, kidney or heart failure, significant heart, lung, digestive, hormone or mental disease or Vitamin B deficiency
* Patients with previous severe head injury or blood clot in the brain
* Patients who are hospitalized, living in nursing homes or residential care facilities
* Patients with brain infections such as abscess, meningitis, encephalitis
* Patients with a history of drug or alcohol abuse

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2001-08; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Time to worsening of symptoms, defined as the time from the beginning of the double-blind portion of the study to the time of an increase in ADAS-cog score of > or = to 4 points

SECONDARY OUTCOMES:
Change in ADAS-cog, CIBIC-plus and DAD scores over time; Safety parameters assessed by adverse events; laboratory tests, vital signs, weight and ECGs.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.p.A. Clinical Trial, Study Director — Janssen-Cilag S.p.A.